CLINICAL TRIAL: NCT02797405
Title: Evaluation of Individual Radiosensitivity of Cancer Patients to be Treated by Radiotherapy or Radiochemotherapy Per-operative
Brief Title: Tumour and HEalthy Tissues DOse-response and Radiosensitivity Assay
Acronym: THEODORA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawal of analysis study Partner.
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ET15-003; 2015-A00931-48 (Other: ID-RCB)
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Sarcoma; Rectal Carcinoma; Esophagus Cancer
Keywords: radiation therapy; radiosensitivity; in vitro diagnostic medical devices; Adverse Event post radiotherapy
MeSH Terms: conditions — Sarcoma; Rectal Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standard treatment (Other): The patients will receive standard treatment according to international recommendations depending on their type of cancer.
  Interventions: Radiation: Standard treatment

INTERVENTIONS:
Radiation: Standard treatment — Sarcoma patients will undergo radiotherapy followed by surgery Rectum cancer patients will undergo radio-chemotherapy followed by surgery Esophagus cancer patients will undergo radio-chemotherapy followed by surgery

SUMMARY:
THEODORA is a prospective pilot clinical trial aiming at first to evaluate and validate the predictive value of the A & MS bioassays on tumor control by radiotherapy.

DETAILED DESCRIPTION:
For that purpose, this project is composed of 3 stages:

* A Calibration stage that will allow to evaluate the correlation between the clinical tumor response parameters (i.e. TV/AP features) and the radiobiological parameters issued from the A/MS bioassays in order to develop a mathematic model defining the UTCR parameter
* A Validation stage in order to assess the validity of A/MS bioassays towards clinical tumour response parameters (i.e. both TV/AP features and UTCR).
* A Precision stage will be performed either to improve the precision of the predictive performance of the A and MS bioassays or to establish a new mathematical model describing the correlation between clinical and radiobiological parameters. The objective of this precision stage will depend of the results of the calibration stage (see below).

This prospective clinical study will be conducted in a population of patients with different tumor types in order to explore a large range of tumor radiosensitivity including sarcomas, rectal carcinoma and esophagus tumor.

ELIGIBILITY:
Inclusion Criteria:

I1. Patients (male or female) ≥ 18 years of age. I2. Adult patients with a suspected, non-treated, non-metastatic retroperitoneal or limb soft tissue sarcoma, esophagus cancer or rectum cancer to be treated by pre-operative radiotherapy or radio-chemotherapy I3. At least one measurable lesion as per RECIST 1.1 I4. Documented negative serology tests (HVB, HIV, HVC) I5. PS ECOG 0 to 1 I6. Patient able and willing to provide informed consent. I7. Ability to understand and willingness for follow-up visits. I8. Covered by a medical insurance.

Exclusion Criteria:

E1. Contra-indication to radiotherapy E2. Contra-indication to skin biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2016-10; Primary Completion 2019-08-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Calibration of the correlation between the clinical tumor response and the results of A/MS bioassays using tumor samples | 2.5 years (after 100 patients enrolled )
  The calibration stage will be performed using data from the first 40 patients enrolled. All the potential correlations between the clinical and radiobiological parameters will be tested. The links between clinical tumor response parameters and radiobiological parameters derived from MS/A bioassays using tumor samples.
Validation of the correlation between the clinical tumor response and the results of A/MS bioassays using tumor samples | 2.5 years (after 100 patients enrolled )
  The validation stage will be performed using data from the remaining 60 patients enrolled. This stage will assess whether or not the prediction of tumor response derived from the A/MS bioassays fits with the observed tumor response after RT.

SECONDARY OUTCOMES:
Validation of the correlation between the healthy tissue response (i.e. AE reported as per CTCAE v4) and the results of MS/A bioassays using skin biopsies | 2.5 years (after 100 patients enrolled )

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre SUNYACH, MD, Principal Investigator — Centre Leon Berard
Locations (7):
- France (7):
  - Centre Francois Baclesse, Caen
  - Infirmerie Protestante, Caluire-et-Cuire
  - Centre Georges-François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - ICL - Institut de Cancérologie de la Lorraine, Vandœuvre-lès-Nancy
  - Hopital Nord Ouest Villefranche Sur Saone, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delaney G, Jacob S, Featherstone C, Barton M. The role of radiotherapy in cancer treatment: estimating optimal utilization from a review of evidence-based clinical guidelines. Cancer. 2005 Sep 15;104(6):1129-37. doi: 10.1002/cncr.21324. PMID 16080176
- [Background] Bentzen SM, Heeren G, Cottier B, Slotman B, Glimelius B, Lievens Y, van den Bogaert W. Towards evidence-based guidelines for radiotherapy infrastructure and staffing needs in Europe: the ESTRO QUARTS project. Radiother Oncol. 2005 Jun;75(3):355-65. doi: 10.1016/j.radonc.2004.12.007. Epub 2005 Mar 16. PMID 16086915
- [Background] Lievens Y, Grau C. Health economics in radiation oncology: introducing the ESTRO HERO project. Radiother Oncol. 2012 Apr;103(1):109-12. doi: 10.1016/j.radonc.2011.12.026. Epub 2012 Feb 8. PMID 22325993
- [Background] Dorr W, Hendry JH. Consequential late effects in normal tissues. Radiother Oncol. 2001 Dec;61(3):223-31. doi: 10.1016/s0167-8140(01)00429-7. PMID 11730991
- [Background] Bodgi L, Granzotto A, Devic C, Vogin G, Lesne A, Bottollier-Depois JF, Victor JM, Maalouf M, Fares G, Foray N. A single formula to describe radiation-induced protein relocalization: towards a mathematical definition of individual radiosensitivity. J Theor Biol. 2013 Sep 21;333:135-45. doi: 10.1016/j.jtbi.2013.05.020. Epub 2013 Jun 2. PMID 23735818
- [Background] Foray N, Colin C, Bourguignon M. 100 years of individual radiosensitivity: how we have forgotten the evidence. Radiology. 2012 Sep;264(3):627-31. doi: 10.1148/radiol.12112560. No abstract available. PMID 22919036
- [Background] Joubert A, Zimmerman KM, Bencokova Z, Gastaldo J, Chavaudra N, Favaudon V, Arlett CF, Foray N. DNA double-strand break repair defects in syndromes associated with acute radiation response: at least two different assays to predict intrinsic radiosensitivity? Int J Radiat Biol. 2008 Feb;84(2):107-25. doi: 10.1080/09553000701797039. PMID 18246480
- [Background] Granzotto A, Joubert A, Viau M, Devic C, Maalouf M, Thomas C, Vogin G, Malek K, Colin C, Balosso J, Foray N. [Individual response to ionising radiation: What predictive assay(s) to choose?]. C R Biol. 2011 Feb;334(2):140-57. doi: 10.1016/j.crvi.2010.12.018. French. PMID 21333944
- [Background] Rothkamm K, Lobrich M. Evidence for a lack of DNA double-strand break repair in human cells exposed to very low x-ray doses. Proc Natl Acad Sci U S A. 2003 Apr 29;100(9):5057-62. doi: 10.1073/pnas.0830918100. Epub 2003 Apr 4. PMID 12679524
- [Background] COPERNIC project investigators; Granzotto A, Benadjaoud MA, Vogin G, Devic C, Ferlazzo ML, Bodgi L, Pereira S, Sonzogni L, Forcheron F, Viau M, Etaix A, Malek K, Mengue-Bindjeme L, Escoffier C, Rouvet I, Zabot MT, Joubert A, Vincent A, Dalla Venezia N, Bourguignon M, Canat EP, d'Hombres A, Thebaud E, Orbach D, Stoppa-Lyonnet D, Radji A, Dore E, Pointreau Y, Bourgier C, Leblond P, Defachelles AS, Lervat C, Guey S, Feuvret L, Gilsoul F, Berger C, Moncharmont C, de Laroche G, Moreau-Claeys MV, Chavaudra N, Combemale P, Biston MC, Malet C, Martel-Lafay I, Laude C, Hau-Desbat NH, Zioueche A, Tanguy R, Sunyach MP, Racadot S, Pommier P, Claude L, Baleydier F, Fleury B, de Crevoisier R, Simon JM, Verrelle P, Peiffert D, Belkacemi Y, Bourhis J, Lartigau E, Carrie C, De Vathaire F, Eschwege F, Puisieux A, Lagrange JL, Balosso J, Foray N. Influence of Nucleoshuttling of the ATM Protein in the Healthy Tissues Response to Radiation Therapy: Toward a Molecular Classification of Human Radiosensitivity. Int J Radiat Oncol Biol Phys. 2016 Mar 1;94(3):450-60. doi: 10.1016/j.ijrobp.2015.11.013. Epub 2015 Nov 14. PMID 26867874
- [Background] Bodgi L, Foray N. The nucleo-shuttling of the ATM protein as a basis for a novel theory of radiation response: resolution of the linear-quadratic model. Int J Radiat Biol. 2016;92(3):117-31. doi: 10.3109/09553002.2016.1135260. PMID 26907628
- [Background] Zaider M, Minerbo GN. Tumour control probability: a formulation applicable to any temporal protocol of dose delivery. Phys Med Biol. 2000 Feb;45(2):279-93. doi: 10.1088/0031-9155/45/2/303. PMID 10701504
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Gerard A, Buyse M, Nordlinger B, Loygue J, Pene F, Kempf P, Bosset JF, Gignoux M, Arnaud JP, Desaive C, et al. Preoperative radiotherapy as adjuvant treatment in rectal cancer. Final results of a randomized study of the European Organization for Research and Treatment of Cancer (EORTC). Ann Surg. 1988 Nov;208(5):606-14. doi: 10.1097/00000658-198811000-00011. PMID 3056288
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Fleming FJ, Pahlman L, Monson JR. Neoadjuvant therapy in rectal cancer. Dis Colon Rectum. 2011 Jul;54(7):901-12. doi: 10.1007/DCR.0b013e31820eeb37. PMID 21654259
- [Background] Movsas B, Diratzouian H, Hanlon A, Cooper H, Freedman G, Konski A, Sigurdson E, Hoffman J, Meropol NJ, Weiner LM, Coia L, Lanciano R, Stein J, Kister D, Eisenberg B. Phase II trial of preoperative chemoradiation with a hyperfractionated radiation boost in locally advanced rectal cancer. Am J Clin Oncol. 2006 Oct;29(5):435-41. doi: 10.1097/01.coc.0000227480.41414.f2. PMID 17023775
- [Background] Wagman R, Minsky BD, Cohen AM, Guillem JG, Paty PP. Sphincter preservation in rectal cancer with preoperative radiation therapy and coloanal anastomosis: long term follow-up. Int J Radiat Oncol Biol Phys. 1998 Aug 1;42(1):51-7. doi: 10.1016/s0360-3016(98)00180-1. PMID 9747819
- [Background] Pisters PW, Harrison LB, Leung DH, Woodruff JM, Casper ES, Brennan MF. Long-term results of a prospective randomized trial of adjuvant brachytherapy in soft tissue sarcoma. J Clin Oncol. 1996 Mar;14(3):859-68. doi: 10.1200/JCO.1996.14.3.859. PMID 8622034
- [Background] Yang JC, Chang AE, Baker AR, Sindelar WF, Danforth DN, Topalian SL, DeLaney T, Glatstein E, Steinberg SM, Merino MJ, Rosenberg SA. Randomized prospective study of the benefit of adjuvant radiation therapy in the treatment of soft tissue sarcomas of the extremity. J Clin Oncol. 1998 Jan;16(1):197-203. doi: 10.1200/JCO.1998.16.1.197. PMID 9440743
- [Background] Koshy M, Rich SE, Mohiuddin MM. Improved survival with radiation therapy in high-grade soft tissue sarcomas of the extremities: a SEER analysis. Int J Radiat Oncol Biol Phys. 2010 May 1;77(1):203-9. doi: 10.1016/j.ijrobp.2009.04.051. Epub 2009 Aug 11. PMID 19679403
- [Background] Strander H, Turesson I, Cavallin-Stahl E. A systematic overview of radiation therapy effects in soft tissue sarcomas. Acta Oncol. 2003;42(5-6):516-31. doi: 10.1080/02841860310014732. PMID 14596510
- [Background] Stacchiotti S, Collini P, Messina A, Morosi C, Barisella M, Bertulli R, Piovesan C, Dileo P, Torri V, Gronchi A, Casali PG. High-grade soft-tissue sarcomas: tumor response assessment--pilot study to assess the correlation between radiologic and pathologic response by using RECIST and Choi criteria. Radiology. 2009 May;251(2):447-56. doi: 10.1148/radiol.2512081403. Epub 2009 Mar 4. PMID 19261927
- [Background] Stahl R, Wang T, Lindner LH, Abdel-Rahman S, Santl M, Reiser MF, Issels RD. Comparison of radiological and pathohistological response to neoadjuvant chemotherapy combined with regional hyperthermia (RHT) and study of response dependence on the applied thermal parameters in patients with soft tissue sarcomas (STS). Int J Hyperthermia. 2009 Jun;25(4):289-98. doi: 10.1080/02656730902873616. PMID 19670096
- [Background] O'Sullivan B, Davis AM, Turcotte R, Bell R, Catton C, Chabot P, Wunder J, Kandel R, Goddard K, Sadura A, Pater J, Zee B. Preoperative versus postoperative radiotherapy in soft-tissue sarcoma of the limbs: a randomised trial. Lancet. 2002 Jun 29;359(9325):2235-41. doi: 10.1016/S0140-6736(02)09292-9. PMID 12103287
- [Background] Cooper JS, Guo MD, Herskovic A, Macdonald JS, Martenson JA Jr, Al-Sarraf M, Byhardt R, Russell AH, Beitler JJ, Spencer S, Asbell SO, Graham MV, Leichman LL. Chemoradiotherapy of locally advanced esophageal cancer: long-term follow-up of a prospective randomized trial (RTOG 85-01). Radiation Therapy Oncology Group. JAMA. 1999 May 5;281(17):1623-7. doi: 10.1001/jama.281.17.1623. PMID 10235156
- [Background] Ishikura S, Nihei K, Ohtsu A, Boku N, Hironaka S, Mera K, Muto M, Ogino T, Yoshida S. Long-term toxicity after definitive chemoradiotherapy for squamous cell carcinoma of the thoracic esophagus. J Clin Oncol. 2003 Jul 15;21(14):2697-702. doi: 10.1200/JCO.2003.03.055. PMID 12860946
- [Background] Morota M, Gomi K, Kozuka T, Chin K, Matsuura M, Oguchi M, Ito H, Yamashita T. Late toxicity after definitive concurrent chemoradiotherapy for thoracic esophageal carcinoma. Int J Radiat Oncol Biol Phys. 2009 Sep 1;75(1):122-8. doi: 10.1016/j.ijrobp.2008.10.075. Epub 2009 Mar 26. PMID 19327900
- [Background] Wahl RL, Jacene H, Kasamon Y, Lodge MA. From RECIST to PERCIST: Evolving Considerations for PET response criteria in solid tumors. J Nucl Med. 2009 May;50 Suppl 1(Suppl 1):122S-50S. doi: 10.2967/jnumed.108.057307. PMID 19403881